CLINICAL TRIAL: NCT00002813
Title: A LIMITED ACCESS PHASE II TRIAL OF CISPLATIN AND NAVELBINE (VINORELBINE) IN ADVANCED AND RECURRENT SQUAMOUS CELL CARCINOMA OF THE CERVIX
Brief Title: Combination Chemotherapy in Treating Patients With Recurrent or Refractory Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000064956; GOG-76Z
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2008-03

CONDITIONS: Cervical Cancer
Keywords: recurrent cervical cancer; stage IVB cervical cancer; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Vinorelbine

INTERVENTIONS:
Drug: cisplatin
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy with cisplatin and vinorelbine in treating patients with refractory or recurrent squamous cell cervical cancer that has not responded to local therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the activity of cisplatin and vinorelbine in terms of response rate, duration of response, time to treatment failure, and survival in patients with advanced, persistent, or recurrent squamous cell carcinoma of the cervix.

OUTLINE: This is a multicenter study. Patients receive vinorelbine IV over 6-10 minutes on days 1, 8, 15, and 22 and cisplatin IV over 4 hours beginning after completion of vinorelbine infusion on day 1. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 28-62 patients will be accrued for this study within approximately 20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced, persistent, or recurrent squamous cell carcinoma of the cervix that failed local therapy and is considered incurable Bidimensionally measurable abdominal, pelvic, or other lesion by palpation, x- ray, or ultrasound If sole site of measurable disease previously irradiated, then documented disease progression at that site required

PATIENT CHARACTERISTICS: Age: Any age Performance status: GOG 0-2 Karnofsky 60%-100% Hematopoietic: WBC at least 3,000/mm3 Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal SGOT no greater than 3 times normal Alkaline phosphatase no greater than 3 times normal Renal: Creatinine no greater than 1.4 mg/dL Creatinine clearance at least 50 mL/min if creatinine greater than 1.2 mg/dL Other: No clinically significant infection No preexisting, clinically significant peripheral neuropathy unless due to cancer No other prior or concurrent malignancy except nonmelanomatous skin cancer No psychological, familial, sociological, or geographical condition that would preclude compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy except for radiosensitization Endocrine therapy: Not specified Radiotherapy: See Chemotherapy Recovered from the toxic effects of any recent radiotherapy Surgery: Recovered from the toxic effects of any recent surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 1997-08; Primary Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Morris, MD, Study Chair — M.D. Anderson Cancer Center
Locations (9):
- United States (9):
  - Chao Family Comprehensive Cancer Center, Orange, California
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Cancer Center of Albany Medical Center, Albany, New York
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brookview Research, Inc., Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Morris M, Blessing JA, Monk BJ, McGehee R, Moore DH. Phase II study of cisplatin and vinorelbine in squamous cell carcinoma of the cervix: a gynecologic oncology group study. J Clin Oncol. 2004 Aug 15;22(16):3340-4. doi: 10.1200/JCO.2004.12.006. PMID 15310778